CLINICAL TRIAL: NCT06885138
Title: Study of the Clinical and Neurophysiological Effects of Transcranial Direct Current Stimulation on Depressive Symptoms in Parkinson's Disease.
Brief Title: Clinical and Neurophysiological Effects of tDCS on Depression in Parkinson's Disease
Acronym: tDCS&PD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4531; tDCS&PD (Other: Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico)
Record Dates: First submitted 2025-02-18; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Depression; Parkinson Disease; tDCS
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham tDCS (Sham Comparator): Patients in this group will receive sham transcranial Direct Current Stimulation (tDCS)
  Interventions: Device: sham transcranial Direct Current Stimulation
- Active tDCS (Experimental): Patients in this group will receive active transcranial Direct Current Stimulation (tDCS) (stimulation polarity: anodal).
  Interventions: Device: active transcranial Direct Current Stimulation

INTERVENTIONS:
Device: active transcranial Direct Current Stimulation — Patients will undergo repeated sessions of active transcranial Direct Current Stimulation (tDCS) (anodal polarity). The active electrode (35 cm²) will be placed over the left dorsolateral prefrontal cortex (DLPFC), while the reference electrode (35 cm²) will be positioned over the contralateral area, with a stimulation intensity of 2mA.
  Patients will undergo a tDCS session on days 1, 2, 3, 4, 5, 12, 19, and 26 of the study. Each session will last 20 minutes.
  Other Names: Neuromodulation
  Arms: Active tDCS
Device: sham transcranial Direct Current Stimulation — Patients will undergo repeated sessions of "sham tDCS." The electrodes will be placed over the left DLPFC and the contralateral area, as in the active stimulation condition. However, the current will be delivered only for the first 5 seconds, preventing the participants from detecting the placebo condition while ensuring that no neuromodulation occurs in the underlying brain areas. Patients will undergo a tDCS session on days 1, 2, 3, 4, 5, 12, 19, and 26 of the study. Each session will last 20 minutes.
  Other Names: Neuromodulation
  Arms: Sham tDCS

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder, characterized by dopaminergic cell degeneration leading to neurophysiological alterations and a heterogeneous clinical presentation. In addition to motor symptoms, PD patients often experience non-motor symptoms, particularly neuropsychiatric manifestations such as depression, anxiety, and apathy. Depression is one of the most prevalent behavioral symptoms, affecting at least 50% of PD patients, with a higher incidence compared to the general population and other disabling conditions. Two main hypotheses explain the emergence of depressive symptoms: one considers depression a reactive response to progressive disability, while the other links it to the underlying neurobiological mechanisms of PD. Additionally, depression and anxiety frequently co-occur in PD, suggesting shared neurobiological pathways.

Conventional pharmacological treatments only partially address affective symptoms in PD, highlighting the need for innovative non-pharmacological therapies. Transcranial direct current stimulation (tDCS) has gained attention as a potential treatment, showing promising results in improving both motor and affective symptoms in PD. While preliminary studies suggest that tDCS may significantly reduce depressive symptoms, current evidence is insufficient to establish clinical recommendations, necessitating further large-scale, randomized controlled trials.

Objectives

The primary objective of this study is to evaluate the effects of repeated tDCS sessions on depressive symptoms in PD patients. Secondary objectives include:

* Assessing the potential impact of repeated tDCS sessions on anxiety, apathy, sleep quality, and quality of life in PD patients.
* Investigating the neurophysiological mechanisms underlying depression and the effects induced by tDCS.

Methodology

Eligible patients will be randomly assigned to one of two groups:

1. Experimental Group: Patients will receive repeated sessions of active tDCS (anodal stimulation). The active electrode (35 cm²) will be placed over the left dorsolateral prefrontal cortex (DLPFC), with the reference electrode (35 cm²) on the contralateral area. Stimulation intensity will be set at 2mA, and each session will last 20 minutes.
2. Control Group: Patients will receive sham tDCS sessions. Electrodes will be positioned identically to the active condition, but the current will only be applied for the first 5 seconds to prevent perception of the sham condition while ensuring no neuromodulatory effects. Each session will last 20 minutes.

Both groups will undergo tDCS sessions on days 1, 2, 3, 4, 5, 12, 19, and 26 of the study.

Assessment and Outcome Measures tDCS treatment will be administered in a hospital setting using the Newronika stimulator (CE-certified medical device). The effects on depressive symptoms and neurophysiological mechanisms will be evaluated using validated clinical scales and neurophysiological assessments at multiple time points:

* T0 (Day 1): Baseline assessment before treatment initiation.
* T1 (Day 5): After one week of treatment.
* T5 (Day 33): One week after completing all treatment sessions.
* T6 (Day 54): One month after treatment completion.

This study aims to improve the understanding of tDCS's clinical efficacy and underlying mechanisms in managing affective symptoms in PD. The findings could support the development of evidence-based non-pharmacological interventions for PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease according to the clinical diagnostic criteria of the Movement Disorder Society;
* No dementia (Montreal Cognitive Assessment score ≥ 22/30);
* Presence of depressive symptoms
* Pharmacological treatment for motor symptoms stable for at least 1 month
* Treatment (pharmacological/non-pharmacological) for depressive symptoms stable for at least 3 months.

Exclusion Criteria:

* Patients with a pacemaker, intracranial electrodes, implanted defibrillators, or any other type of prosthesis;
* Patients undergoing Deep Brain Stimulation treatment;
* Patients with epilepsy or a history of seizures;
* Patients with psychosis;
* Patients with a history of skull fracture;
* Pregnant/breastfeeding patients;
* Patients with suicidal ideation or a suicide attempt in the six months prior to the start of the study;
* Patients with a history of substance dependence or abuse;
* Concomitant treatment with medications that may affect tDCS (benzodiazepines, anticonvulsants, pseudoephedrine, dextromethorphan).

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Enrollment: 52 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The Beck Depression Inventory-II (BDI-II) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Each item is scored on a scale from 0 to 3, with total scores ranging from 0 to 63. Higher scores indicate more severe depressive symptoms.
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which mental health professionals use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated from 0 to 6, leading to a total score range of 0 to 60. Higher scores indicate more severe depression.
Visual Analog Scale (VAS) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The Visual Analog Scale (VAS) for mood is a widely used tool to assess a person's emotional state. It consists of a straight line, usually 100 mm in length, with one end representing the most negative mood state (e.g., very sad, depressed) and the other end representing the most positive mood state (e.g., very happy, elated). The individual marks a point on the line that corresponds to their current mood, and the distance from the "negative" end to the mark is then measured in millimeters, providing a quantitative measure of the individual's emotional state. Scores range from 0 to 10, with higher scores indicating a more positive mood. This scale is easy to use and provides a subjective yet reliable way to track mood changes over time.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Total scores range from 20 to 80 for each subscale, with higher scores indicating greater anxiety.
Apathy Evaluation Scale (AES) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The Apathy Evaluation Scale (AES) is a 18-item self-report questionnaire assessing apathy in behavioral, cognitive, and emotional domains. Each item is rated on a 4-point Likert scale (1 = not at all, 4 = a lot). Total scores range from 18 to 72, with higher scores indicating greater levels of apathy.
Parkinson's Disease Questionnaire-8 (PDQ-8) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The Parkinson's Disease Questionnaire-8 (PDQ-8) is a self-report measure derived from the PDQ-39. It assesses health-related quality of life in individuals with Parkinson's disease across eight key domains, providing a brief yet effective evaluation of disease impact. It consists of 8 items, each rated on a 5-point Likert scale (0 = never, 4 = always). The total score is transformed to a 0-100 scale, where higher scores indicate worse health-related quality of life.
Pittsburgh Sleep Quality Index (PSQI) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report questionnaire assessing sleep quality over the past month. It evaluates seven components (e.g., sleep duration, disturbances, latency, and daytime dysfunction), each scored from 0 to 3, yielding a global score ranging from 0 to 21. Higher scores indicate poorer sleep quality
EEG Peak Frequency in the Beta Band (Hz) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The EEG peak frequency in the beta band (13-30 Hz) reflects cortical activity associated with cognitive processing, alertness, arousal, and emotional regulation. Changes in peak beta frequency may indicate alterations in neurophysiological functioning. Higher values are generally linked to increased cortical activation, while lower values may reflect reduced cortical excitability.
Blink Reflex Area (mV·ms) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The blink reflex (BR) area quantifies the overall amplitude of the reflexive eye closure response to external stimuli. It provides information about brainstem excitability and neuromuscular response intensity.
Blink Reflex Duration (ms) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The blink reflex (BR) duration represents the total time from the initiation to the completion of the reflexive eye closure. Prolonged duration may reflect altered neural conduction or motor control.
Blink Reflex Latency (ms) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The blink reflex (BR) latency is the time interval between the stimulus and the onset of the eye closure response. It serves as an indicator of neural transmission efficiency within the trigeminal-facial circuitry.
Startle Saccadic Reflex Area (mV·ms) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The startle saccadic reflex (SSR) area measures the magnitude of the rapid eye movement response to a sudden stimulus, providing insight into sensorimotor integration and brainstem responsiveness.
Startle Saccadic Reflex Duration (ms) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The startle saccadic reflex (SSR) duration refers to the total time span of the reflexive saccadic eye movement. Prolonged duration may reflect changes in neuromuscular coordination and sensorimotor processing.
Startle Saccadic Reflex Latency (ms) | Baseline (T0); on day 5 (T1); one week after the end of treatment on day 33 (T2); one month after the end of treatment on day 54 (T3)
  The startle saccadic reflex (SSR) latency is the time interval between the presentation of a sudden stimulus and the initiation of the saccadic eye movement. It provides a measure of neural conduction speed in reflex pathways.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No